CLINICAL TRIAL: NCT02089451
Title: A Trial Comparing the Pharmacokinetic Properties of FIAsp After Different Injection Regions and Routes of Administration in Healthy Subjects
Brief Title: A Trial Comparing the Pharmacokinetic Properties of Faster-acting Insulin Aspart (FIAsp) After Different Injection Regions and Routes of Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1218-3949; 2011-002590-32 (EudraCT Number); U1111-1121-8351 (Other: WHO)
Record Dates: First submitted 2014-01-30; First posted 2014-03-17 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FIAsp (Experimental): Each subject will be randomised to a treatment sequence consisting of 5 treatment periods
  Interventions: Drug: Faster-acting insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Drug: insulin aspart (faster acting insulin aspart) Subjects will receive five single dose level of faster acting insulin aspart. Three single dose s.c under the skin (abdomen, deltoid/upper arm, thigh), one single dose i.m. (intramuscularly, into the muscle) and one single dose i.v. (intravenously, into the vein)

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to compare the pharmacokinetic properties (the exposure of the trial drug in the body) of faster-acting insulin aspart (FIAsp) after different injection regions and routes of administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years both inclusive at the time of signing informed consent
* Considered generally healthy upon completion of medical history, physical examination,analysis of laboratory safety variables, vital signs and ECG (electrocardiogram), as judged by the investigator
* Body mass index 20.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve (only for subcutaneous administration) | From 0 to 12 hours

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve (only for intramuscular administration) | From 0 to 12 hours
Maximum observed serum insulin aspart concentration (only for subcutaneous and intramuscular administration) | From 0 to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Hovelmann U, Heise T, Nosek L, Sassenfeld B, Thomsen KMD, Haahr H. Pharmacokinetic Properties of Fast-Acting Insulin Aspart Administered in Different Subcutaneous Injection Regions. Clin Drug Investig. 2017 May;37(5):503-509. doi: 10.1007/s40261-017-0499-y. PMID 28185141
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com